CLINICAL TRIAL: NCT00364806
Title: Prochlorperazine Verus Metoclopramide for the Treatment of Acute Migraine in the Emergency Department Setting
Brief Title: Prochlorperazine vs Metoclopramide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Prof. Emergency Medicine, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-06-311
Record Dates: First submitted 2006-08-14; First posted 2006-08-16 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Migraine
Keywords: Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Prochlorperazine; Metoclopramide

INTERVENTIONS:
Drug: Prochlorperazine
Drug: Metoclopramide

SUMMARY:
Migraine headaches are a common reason for patients to present to an emergency department. We are comparing two different medications to see which one is better for patients who present ot an emergency room with a migraine headache.

DETAILED DESCRIPTION:
One-third of the five million headache patients who present to US Emergency Departments (ED) annually have a migraine headache. The anti-emetic dopamine receptor antagonists have proven efficacy for migraines, are at least as well-tolerated as triptans, and enjoy wide-spread use in North American EDs. However, it is not yet clear which medication within this class and which dosage is optimal. Therefore, we propose a randomized clinical trial to compare the efficacy and tolerability of two standard medications for migraine.

Specific Aim: To compare the efficacy of metoclopramide versus prochlorperazine for the emergency department treatment of migraine headaches. Both of these medications will be combined with diphenhydramine to prevent extra-pyramidal side effects.

Patients will be enrolled as participants if they present to one of the participating EDs and consent to participate. Medications will be administered as an intravenous drip over 15 minutes. Rescue medication will be administered, if needed, after one hour. A follow-up phone call will be conducted 24 hours after the ED visit.

ELIGIBILITY:
Inclusion Criteria:

* Present to the Ed with an acute migraine headache

Exclusion Criteria:

* secondary headache
* if the patient is to receive a lumbar puncture in the ED
* maximum temperature greater than 100.3 degrees
* new objective neurologic abnormality at the time of physical exam
* allergy or intolerance to a study medication
* pregnancy
* previous enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76
Dates: Start 2006-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
One hour pain scores

SECONDARY OUTCOMES:
One hour, two hour and 24 hour pain, functional disability scores, and side effect profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Friedman, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States